CLINICAL TRIAL: NCT03583723
Title: Adaptive Radiation Therapy in Locally Advanced Non-Small Cell Lung Cancer (LARTIA Trial)
Brief Title: Adaptive Radiotherapy in Locally Advanced Non-Small Cell Lung Cancer (LARTIA Trial)
Acronym: LARTIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Michele Fiore, Researcher, Medical Doctor, Campus Bio-Medico University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60/12 PAR ComEt CBM
Record Dates: First submitted 2018-06-27; First posted 2018-07-11 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Adaptive radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy Group (Experimental): Patients with LA NSCLC treated with concurrent chemoradiation will be enrolled. During treatment all patients will undergo weekly chest CT simulations without intravenous contrast to assess acute toxicity and tumor shrinkage, and they will be all visualized by two radiation oncologists independently. For all CT simulations, each physician will be able to judge whether reduction will be (1) present and clinically significant, (2) present and clinically non significant, or (3) absent. In the case of physician agreement for the first category, a contrast-enhanced CT will be performed to better visualize node reduction, a new target volume will be delineated, and a new treatment plan (replanning study) performed. Patients will be treated without any time break.
  Interventions: Radiation: Radiotherapy Group

INTERVENTIONS:
Radiation: Radiotherapy Group — Patients will be immobilized with customized devices. Either four-dimensional CT or slow CT images using a multislice CT scanner will be acquired to evaluate internal target motion. Initially, gross tumor volume (GTV) will be determined in the maximum intensity projection on the initial size of the tumor and involved lymph nodal sites defined as PET-positive nodes and/or a node diameter greater than 1 cm, clinical target volume (CTV) will be defined as equal to the GTV plus node-positive stations and hilar stations, and planning target volume (PTV) will be created equal to the CTV plus a 0.5-cm safety margin. Treatment will be performed with a linear accelerator in a photon regimen, with a 6-to 15-megavolt (MV) nominal energy and three-dimensional (3D) conformal technique.

SUMMARY:
Anatomical change of tumor during radiotherapy contributes to target missing. However, in the case of tumor shrinkage, adaptation of volume could result in an increased incidence of recurrence in the area of target reduction. This study aims to investigate the incidence of failure of the adaptive approach in Locally Advanced Non-Small Cell Lung Cancer and, in particular, the risk for local recurrence in the area excluded after replanning.

DETAILED DESCRIPTION:
Concurrent chemoradiation is the standard of care for patients affected by locally advanced (LA) NSCLC. Its superiority over radiotherapy alone or sequential chemoradiation has been proved in multiple phase III randomized trials. In a meta-analysis of six randomized studies, concurrent chemoradiotherapy decreased locoregional progression by 6.1% at 5 years when compared with sequential chemoradiation. This resulted in an improvement in overall survival of 4.5% at 5 years that was possibly directly related to locoregional control. Many patients however succumb to locoregional failure or distant metastases. Thanks to modern radiotherapy techniques, some strategies manage the geometrical uncertainties of imaging, treatment planning, and treatment delivery and thereby improve target coverage with a much steeper dose gradient and less irradiated normal tissue. The introduction of image-guided radiotherapy reveals the occurrence of target changes during treatment, and although the percentage of patients who experienced regression is not high (range 25%-40%), the degree of regression is in the range of 29% to 40%, corresponding to a rate of tumor shrinkage per fraction of 0.79% to 1.65%. Anatomical changes during radiotherapy might introduce discrepancies between the planned and delivered dose. Currently, the literature reports only dosimetric experiences and lacks clinical data on outcome when patients are treated with the adaptive approach. This study aims to investigate the failure pattern in patients with LA NSCLC treated with concurrent chemoradiotherapy with an adaptive approach, in particular, to evaluate the risk for local recurrence in the area excluded during replanning.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven NSCLC;
* inoperable stage IIIA/IIIB disease and intrathoracic relapse after surgery;
* positron emission tomography (PET)/computed tomography (CT) and/or total-body CT with contrast excluding metastatic disease (including brain);
* no previous radiotherapy treatment;
* Eastern Cooperative Oncology Group performance status of 0 to 1;
* clinically measurable/evaluable disease;
* minimum life expectancy of 12 weeks;
* adequate respiratory, renal, hepatic and bone marrow function and non-contraindicative cardiovascular disease.

Exclusion Criteria:

* previous radiotherapy treatment
* concurrent systemic disorders incompatible with chemotherapy or radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11-02 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2019-01-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Local Recurrence and Pattern of Failure | three months
  Patients are not considered to have local-regional control unless they achieve at least a partial response of their primary tumor or stable disease by imaging. Patients who do not achieve objective response are considered to have local-regional failure. Local-regional control rates are analyzed using the Kaplan-Meier method. Local recurrences are defined according to a dimensional and metabolic increase at chest CT with intravenous contrast and fludeoxyglucose F 18 (FDG) PET/CT. Recurrences are identified visually and independently by three radiation oncologists with the same method. The modality for definition of failures is readjusted with these definitions: "in-field failure" when a dimensional and/or metabolic progression is reported within the replanning PTV; "marginal failure" in cases of recurrence in the initial PTV but not in the replanning PTV, and "out-of-field failure" if the recurrence occurs outside the initial PTV.

SECONDARY OUTCOMES:
Response evaluation | three months
  Response evaluation is defined according to the Response Evaluation Criteria in Solid Tumors criteria for complete and partial response, progression, and stable disease.
Overall Survival | three years
  Overall Survival is determined from the day of the diagnosis to the death, or to the last follow-up if no event is observed
Progression-Free Survival | three years
  Progression-free survival is obtained from the beginning of treatment to the observation of progression/recurrence, or to the last follow-up if no event is observed.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ramella, Prof, Study Director — Campus Bio-Medico University
Locations (1):
- Michele Fiore, Rome, Italy

IPD SHARING:
Plan to Share IPD: No